CLINICAL TRIAL: NCT05944289
Title: Acceptance and Commitment Therapy for Stress Reduction in Caregivers of Children With Autism Spectrum Disorder: A Pilot Study
Brief Title: Pilot Study: Stress Reduction in Caregivers of Children With ASD Using ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fielding Graduate University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-0404
Record Dates: First submitted 2023-05-30; First posted 2023-07-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Caregiver Stress
Keywords: Caregivers of children with autism and stress
MeSH Terms: conditions — Caregiver Burden | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to a treatment condition (parent support control group or ACT intervention group). The design of the study will be randomized, two-group mixed model design with 1) a group-based Acceptance and Commitment Therapy (ACT)intervention and 2) a parent support group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT (Experimental): ACT Intervention Group
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Support (Other): Control Group - Caregiver support group
  Interventions: Behavioral: Caregiver Support Group

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — a four-week workshop based on the principles and procedures of Acceptance and Commitment Therapy
  Arms: ACT
Behavioral: Caregiver Support Group — Caregiver support group to run parallel to the ACT intervention group.
  Arms: Support

SUMMARY:
Parents/Caregivers of children with autism need psychological flexibility and self-efficacy for the ACT program to be effective.

This study will compare intervention differences between groups. Repeated measures will be given three times (pre-intervention, post-intervention, and follow-up) to an ACT intervention group and a support group (control). The purpose of the present study is to compare the effects of a brief ACT-based workshop for parents of children with autism with a concurrent parent support control group using a variety of self-report measures addressing psychological flexibility, depression, thought suppression, cognitive fusion, positive aspects of caregiving, stress, self-compassion, and valued living.

ELIGIBILITY:
Inclusion Criteria:

* Individuals will be eligible for entry if (1) they are the biological or adoptive parent (and primary caregiver) of a child with a diagnosis of an autism spectrum disorder, (2) the child is 2-17 years of age inclusive, (3) speak English, and (4) they plan to live in the area for at least six months and (5) present proof of vaccination and (6) agree to masking and social distancing during the in-person workshop.

Exclusion Criteria:

* Individuals will be excluded from the study if (1) they are involved in a concurrent clinical trial of psychosocial interventions for parents/caregivers or (2) they (or their child/spouse) indicate during telephone screening or on the demographics questionnaire active major medical issues such as cancer, organ transplant, or severe mental health disorders that prevent active participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-19 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
Brief Symptom Inventory-18 (BSI-18) | Baseline - prior to intervention particpation
  18-item self-administered measure that provides information on participants' overall psychological distress and Global Severity Index, as well as scales of somatization, depression, and anxiety
Brief Symptom Inventory-18 (BSI-18) | Post - within two weeks of intervention completion
  18-item self-administered measure that provides information on participants' overall psychological distress and Global Severity Index, as well as scales of somatization, depression, and anxiety
Brief Symptom Inventory-18 (BSI-18) | Follow-up- completed within 1 month of intervention completion
  18-item self-administered measure that provides information on participants' overall psychological distress and Global Severity Index, as well as scales of somatization, depression, and anxiety
Perceived Stress Scale - 10 Items (PSS-10) | Baseline - prior to intervention particpation
  10-item questionnaire used to measure the degree to which life has been experienced as unpredictable, uncontrollable, and overloaded
Perceived Stress Scale - 10 Items (PSS-10) | Post - within two weeks of intervention completion
  10-item questionnaire used to measure the degree to which life has been experienced as unpredictable, uncontrollable, and overloaded
Perceived Stress Scale - 10 Items (PSS-10) | Follow-up- completed within 1 month of intervention completion
  10-item questionnaire used to measure the degree to which life has been experienced as unpredictable, uncontrollable, and overloaded
Positive Aspects of Caregiving (PAC) | Baseline - prior to intervention particpation
  nine-item pencil-and-paper instrument that assesses caregivers' subjectively perceived gains from desirable aspects of or positive affective returns from providing care for their loved one
Positive Aspects of Caregiving (PAC) | Post - within two weeks of intervention completion
  nine-item pencil-and-paper instrument that assesses caregivers' subjectively perceived gains from desirable aspects of or positive affective returns from providing care for their loved one
Positive Aspects of Caregiving (PAC) | Follow-up- completed within 1 month of intervention completion
  nine-item pencil-and-paper instrument that assesses caregivers' subjectively perceived gains from desirable aspects of or positive affective returns from providing care for their loved one
Parental Stress Index-Short Form (PSI-SF) | Baseline - prior to intervention particpation
  36-item self-report instrument
Parental Stress Index-Short Form (PSI-SF) | Post - within two weeks of intervention completion
  36-item self-report instrument
Parental Stress Index-Short Form (PSI-SF) | Follow-up- completed within 1 month of intervention completion
  36-item self-report instrument
Self-Compassion Scale - Short Form (SCS-SF) | Baseline - prior to intervention particpation
  12-item self-report measure of self-compassion, such as self-kindness, self-judgment, common humanity, isolation, mindfulness, and overidentification
Self-Compassion Scale - Short Form (SCS-SF) | Post - within two weeks of intervention completion
  12-item self-report measure of self-compassion, such as self-kindness, self-judgment, common humanity, isolation, mindfulness, and overidentification
Self-Compassion Scale - Short Form (SCS-SF) | Follow-up- completed within 1 month of intervention completion
  12-item self-report measure of self-compassion, such as self-kindness, self-judgment, common humanity, isolation, mindfulness, and overidentification

CONTACTS AND LOCATIONS:
Overall Officials: Asimina Lazaridou, Ph.D, Study Chair — Fielding Graduate University
Locations (1):
- Fielding Graduate University, Santa Barbara, California, United States

IPD SHARING:
Plan to Share IPD: No
In the following standard research practices, the data will never contain identifying or potentially identifying information. The participant identities and responses to assessments will be downloaded from Qualtrics and stored only on Shannon Harper's password-protected computer. The data will be saved on a password-protected computer for 10 years after publication, and then the data will be destroyed.